CLINICAL TRIAL: NCT01574053
Title: Enroll -HD: A Prospective Registry Study in a Global Huntington's Disease Cohort
Status: Recruiting | Type: Observational
Sponsor: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Enroll -HD
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; Huntington Disease; Juvenile Huntington's Disease; Registry; Cohort; CHDI
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Enroll-HD is a longitudinal, observational, multinational study that integrates two former Huntington's disease (HD) registries-REGISTRY in Europe, and COHORT in North America and Australasia-while also expanding to include sites in Latin America. More than 30,000 participants have now enrolled into the study. With annual assessments and no end date, Enroll-HD has built a large and rich database of longitudinal clinical data and biospecimens that form the basis for studies developing tools and biomarkers for progression and prognosis, identifying clinically-relevant phenotypic characteristics, and establishing clearly defined endpoints for interventional studies. Periodic cuts of the database are now available to any interested researcher to use in their research - visit www.enroll-hd.org/for-researchers/access-data/ to learn more.

DETAILED DESCRIPTION:
The primary objective of Enroll-HD is to develop a comprehensive repository of prospective and systematically collected clinical research data (demography, clinical features, family history, genetic characteristics) and biological specimens (blood) from individuals with manifest HD, unaffected individuals known to carry the HD mutation or at risk of carrying the HD mutation, and control research participants (e.g., spouses, siblings or offspring of HD mutation carriers known not to carry the HD mutation). Enroll-HD is conceived as a broad-based and long-term project to maximize the efficiencies of non-clinical research and participation in clinical research. With more than 150 active clinical sites in 23 countries, Enroll-HD is now the largest HD database available and is accessible to any interested researcher - visit www.enroll-hd.org/for-researchers/access-data/ to learn more.

ELIGIBILITY:
Inclusion Criteria:

* Carriers: This group comprises the primary study population and consists of individuals who carry the HD gene expansion mutation.
* Controls: This group comprises the comparator study population and consists of individuals who do not carry the HD expansion mutation.

These two major categories can be further subdivided into six different subgroups of eligible individuals:

* Manifest/Motor-manifest HD: Carriers with clinical features that are regarded in the opinion of the investigator as diagnostic of HD.
* Pre-Manifest/-Motor-manifest HD: Carriers without clinical features regarded as diagnostic of HD.
* Genotype Unknown: This group includes a first or second degree relative (i.e., related by blood to a carrier) who has not undergone predictive testing for HD and therefore has an undetermined carrier status.
* Genotype Negative: This group includes a first or second degree relative (i.e., related by blood to a carrier) who has undergone predictive testing for HD and is known not to carry the HD expansion mutation.
* Family Control: Family members or individuals not related by blood to carriers (e.g., spouses, partners, caregivers).
* Community Controls: Individuals unrelated to HD carriers who did not grow up in a family affected by HD. Data collected from community controls will be used for generation of normative data for sub-studies.

Participant status will be captured in the study database using 2 variables: 1) Investigator Determined Status: this will be based on clinical signs and symptoms and genotyping performed as part of medical care, and will be updated at every visit; and 2) Research Genotyping Status: this will be based on genotyping conducted as part of Enroll-HD study procedures. Based on research genotyping, participants will be reclassified under this variable from Genotype Unknown to 'Carriers' or 'Controls'. Investigators and participants will be blinded to this reclassification.

Exclusion Criteria:

* Individuals who do not meet inclusion criteria,
* Individuals with choreic movement disorders in the context of a negative test for the HD gene mutation.
* For Community Controls: those individuals with a major central nervous system disorder will be excluded (e.g. stroke, Parkinson's disease, multiple sclerosis, etc.).

Participants under 18 may be eligible to participate (if they have juvenile-onset HD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with HD and their family members are recruited from specialty clinics (Human Genetics, Neurology, Psychiatry) that advise and treat people affected by HD. In addition, in some areas community clinics and neurologists who see HD patients recruit participants for this study. Participants also receive information about the study through websites, clinical practices, support groups, advocacy newsletters, etc. and place a direct request to be considered for participation in the study. Community controls are identified by study site staff (using advertisements, flyers and newsletters) with the support of the Enroll-HD operational staff.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2062-01 (Estimated); Study Completion 2062-01 (Estimated)

PRIMARY OUTCOMES:
Motor Assessments: Unified Huntington's Disease Rating Scale (UHDRS) 99 Motor, UHDRS '99 Diagnostic Confidence Level | through study completion, an average of 1 year
  The motor section of the UHDRS assesses motor features of HD with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural stability. UHDRS 99 Motor, UHDRS Diagnostic Confidence Level.
Functional Assessments: UHDRS '99 Total Functional Capacity, UHDRS '99 Functional Assessment Scale, UHDRS '99 Independence Scale | through study completion, an average of 1 year
  The Total Functional Capacity, Functional Assessment and Independence Subscales of the UHDRS '99 will be used to assess participants' functional status. The Total Functional Capacity scale has established psychometric properties including inter-rater reliability and validity, based on radiographic measures of disease progression.
Problem Behaviors Assessment-Short (PBA-s) | through study completion, an average of 1 year
  The Problem Behavioral Assessment Short Version (PBA-s) will be used to perform behavioral assessments. This instrument measures frequency and severity of symptoms related to altered affect, thought content and coping styles.
Cognitive Assessments: Symbol Digit Modality Test; Stroop Color Naming; Stroop Word Reading; Categorical Verbal Fluency | through study completion, an average of 1 year
  Cognition will be assessed using the Categorical Verbal Fluency Test, Symbol Digit Modality Test and Stroop Color and Word Reading Test. Verbal fluency is a commonly used neuropsychological test which examines the ability to spontaneously produce words orally within a fixed time span. For category fluency, words must be produced according to semantic constraints. The measure of performance used will be the number of correctly generated words within 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard G Landwehrmeyer, MD, PhD, Principal Investigator — University of Ulm; Jamie Levey, Study Director — CHDI Foundation, Inc.
Locations (183):
- United States (62):
  - University of Alabama, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California - Irvine Medical Center, Irvine, California
  - Loma Linda Medical Center, Loma Linda, California
  - University of California - Los Angeles, Los Angeles, California
  - University of California - Davis, Sacramento, California
  - University of California - San Diego, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - Cenexel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida Board of Trustees, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, HDSA Center of Excellence at USF, Tampa, Florida
  - Emory University, Wesley Woods Health Center, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois College of Medicine at Rockford, Rockford, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hereditary Neurological Disease Center, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic - Las Vegas, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers, the State University of New Jersey, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Sanford Health, Fargo, North Dakota
  - University of Cincinatti, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Parkinson's and Movement Disorders Center, Henrico, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Booth Gardner Parkinson's Care Center (Evergreen Health), Kirkland, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Instituto de Neurociencias Buenos Aires (INEBA), Buenos Aires, Argentina
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Monash University, Melbourne, Victoria
  - The Neurosciences Unit - North Metropolitan Hospital, Perth, Western Australia
  - University of Melbourne, Royal Melbourne Hospital, Parkville
- Universitatsklinik Innsbruck, Innsbruck, Austria
- Belgium (4):
  - University Hospitals Leuven, Leuven, Vlaams-Brabant
  - Bruxelles - Erasme, Brussels
  - Institut de Pathologie et de Génétique (IPG), Charleroi
  - Hôpital du Beau Vallon ASBL, Saint-Servais
- Canada (9):
  - University of Calgary, Movement Disorders Program, Calgary, Alberta
  - University of Alberta (Glenrose), Edmonton, Alberta
  - University of Alberta Hospital in Edmonton, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Centre for Movement Disorders, Markham, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - CHUM Hospital of Notre Dame, Montreal, Quebec
- CETRAM, Santiago, Chile
- Colombia (2):
  - Universidad de Antioquia, Grupo de Neurociencias, Medellín, Antioquia
  - Servicios Médicos MS, Clínica de Marly, Bogotá, Cundinamarca
- Denmark (3):
  - University Hospital of Aarhus, Aarhus
  - University Hospital of Copenhagen, Copenhagen
  - University Hospital of Odense, Odense
- France (11):
  - Hôpitaux Universitaires de Strasbourg Hôpital de Hautepierre-Service de Neurologie, Strasbourg, Alsace Lorraine
  - CHU Amiens-Picardie, Amiens
  - CHU Angers, Centre de Référence Maladies Neurogénétiques, Angers
  - Bordeaux - Huntington Disease competencies center, Bordeaux
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - Hôpital Henri Mondor, Centre d'Investigation Clinique, Créteil
  - Lille-Amiens - Huntington Disease Constituent site, Lille
  - Hôpital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - Institut du Cerveau et de la Moelle Epinière, Paris
  - Hôpital Purpan, Centre d'Investigation Clinique, Toulouse
- Germany (14):
  - University Hospital Aachen, Aachen
  - University of Berlin, Berlin
  - St. Josef und St. Elisabeth Hospital, Bochum
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - University Hospital Erlangen, Erlangen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Paracelsus Elena Klinik Kassel, Kassel
  - University Hospital Schleswig-Holstein, Lübeck
  - University Hospital Giessen and Marburg, Marburg
  - Technical University of Munich, Munich
  - George-Huntington-Institut GmbH, Münster
  - kbo-Isar-Amper-Klinikum Taufkirchen (Vils), Taufkirchen
  - University Hopsital of Ulm, Ulm
  - University Hospital of Wuerzburg, Würzburg
- Beaumont Hospital, Dublin, Republic of Ireland, Ireland
- Italy (9):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta - Genetics, Milan, MI
  - Bari Policlinico General Hospital, Bari
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Università degli Studi di Genova (DINOGMI), Genoa
  - Fondazione IRCCS Istituto Neurologico Carlo Besta - Neurology, Milan
  - University of Naples, Napoli
  - Università Cattolica del Sacro Cuore, Rome
  - Lega Italiana Ricerca Huntington (LIRH), Rome
  - Azienda Ospedaliera Sant'Andrea, Rome
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Clinical Trial Center Maastricht B.V., Maastricht
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - New Zealand Brain Research Institute at University of Otago, Christchurch
  - Wellington Hospital, Wellington
- Poland (6):
  - Copernicus Podmiotem Leczniczym sp. z o.o., Gdansk
  - Krakowska Akademia Neurologii Sp. z o.o, Katowice
  - Krakow - Krakowska Akademia Neurologii, Krakow
  - Solumed Centrum Medyczne, Poznan
  - Medical University of Warsaw, Warsaw
  - Institute of Psychiatry and Neurology, Warsaw, Warsaw
- Portugal (5):
  - Hospital Prof Doutor Fernando Fonseca, Amadora
  - Hospital Universitário de Coimbra, Coimbra
  - Central Lisbon Hospital, Lisbon
  - Hospital de Santa Maria / Instituto de Medicina Molecular, Lisbon
  - Hospital Universitário de São João, Porto
- Spain (12):
  - Hospital Infanta Cristina, Badajoz, Badajoz
  - Hospital de Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Mare de Déu de la Mercè, Barcelona
  - Fundacion Clinic per a La Recerca Biomèdica, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Fundacion Hospital Universitario La Fe, Valencia
- Switzerland (2):
  - Siloah AG, Gümligen
  - University Hospital Zurich, Zurich
- United Kingdom (30):
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Leicestershire Partnership, Narborough, Leicestershire
  - North Bristol NHS Trust, Bristol, UK
  - Fife Health Board, Kirkcaldy, UK
  - Betsi Cadwaladr University Health Board, Wrexham, UK
  - University of Aberdeen, Aberdeen
  - Birmingham and Solihull Mental Health NHS Foundation Trust, Birmingham
  - University of Cambridge, Cambridge
  - Cardiff University, Cardiff
  - Tayside Health Board, Dundee
  - Lothian Health Board, Edinburgh
  - Greater Glasgow Health Board, Glasgow
  - Ayrshire Central Hospital, Kilmarnock
  - NHS Forth Valley, Larbert
  - Leeds Teaching Hospitals, Leeds
  - The Walton Centre, Liverpool
  - Guy's and St. Thomas's NHS Foundation Trust, London
  - St. George's Hospital, London
  - University College of London, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Northumberland, Tyne & Wear NHS Foundation Trust of St. Nicholas Hospital, Newcastle upon Tyne
  - St. Andrews Healthcare, Northampton
  - Oxford Radcliffe Hospitals, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - Poole Hospital, Poole
  - Royal Berkshire NHS Foundation Trust, Reading
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - University Hospital Southampton, Southampton
  - North Staffordshire Combined Healthcare NHS Trust, Stoke-on-Trent
  - Avon and Wiltshire Mental Health Partnership, Swindon

REFERENCES:
- [Derived] Gray SM, Dai J, Smith AC, Beckley JT, Rahmati N, Lewis MC, Quirk MC. Changes in 24(S)-Hydroxycholesterol Are Associated with Cognitive Performance in Early Huntington's Disease: Data from the TRACK and ENROLL HD Cohorts. J Huntingtons Dis. 2024 Nov;13(4):449-465. doi: 10.3233/JHD-240030. PMID 39269850
- [Derived] Langbehn DR, Sathe SS, Loy C, Sampaio C, Mccusker EA. A Phenotypic Atlas for Huntington Disease Based on Data From the Enroll-HD Cohort Study. Neurol Genet. 2023 Nov 28;9(6):e200111. doi: 10.1212/NXG.0000000000200111. eCollection 2023 Dec. PMID 38035176
- [Derived] Landwehrmeyer GB, Fitzer-Attas CJ, Giuliano JD, Goncalves N, Anderson KE, Cardoso F, Ferreira JJ, Mestre TA, Stout JC, Sampaio C. Data Analytics from Enroll-HD, a Global Clinical Research Platform for Huntington's Disease. Mov Disord Clin Pract. 2016 Jun 22;4(2):212-224. doi: 10.1002/mdc3.12388. eCollection 2017 Mar-Apr. PMID 30363395